CLINICAL TRIAL: NCT06153355
Title: Single- and Multiple-Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of LY3839840 Following Oral Dosing in Healthy Participants
Brief Title: A First-In-Human Study of LY3839840 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18798; J4U-MC-KTAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part E is non-randomized and open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LY3839840 (Part A) (Experimental): Single ascending dose of LY3839840 administered orally.
  Interventions: Drug: LY3839840
- LY3839840 (Part B) Cohort 1-3 (Experimental): Multiple ascending dose of LY3839840 administered orally.
  Interventions: Drug: LY3839840
- LY3839840 (Part B) Cohort 4 (Experimental): Multiple ascending dose of LY3839840 administered orally.
  Interventions: Drug: LY3839840
- LY3839840 (Part B) Optional Cohort 5 (Experimental): Multiple ascending dose of LY3839840 administered orally pending data from Cohort 4
  Interventions: Drug: LY3839840
- LY3839840 (Part C) (Experimental): Single and multiple dose of LY3839840 administered orally in Chinese participants.
  Interventions: Drug: LY3839840
- LY3839840 (Part D) (Experimental): Multiple ascending dose of LY3839840 administered orally in Japanese participants.
  Interventions: Drug: LY3839840
- Placebo (Parts A-D) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo
- Midazolam (Part E) (Experimental): Midazolam substrate alone or with LY3839840 administered orally
  Interventions: Drug: LY3839840; Drug: Midazolam

INTERVENTIONS:
Drug: LY3839840 — Administered orally.
  Arms: LY3839840 (Part A); LY3839840 (Part B) Cohort 1-3; LY3839840 (Part B) Cohort 4; LY3839840 (Part B) Optional Cohort 5; LY3839840 (Part C); LY3839840 (Part D); Midazolam (Part E)
Drug: Placebo — Administered orally.
  Arms: Placebo (Parts A-D)
Drug: Midazolam — Administered orally
  Arms: Midazolam (Part E)

SUMMARY:
The main purpose of this first-in-human study to investigate the safety of LY3839840 in single and multiple doses, and how it's processed in the body when given in different amounts.

DETAILED DESCRIPTION:
The study will be conducted in five parts (A, B, C, D, and E) and each enrolled participant will receive a single dose (Parts A and C) or multiple dose (Parts B, C and D) of either LY3839840 or placebo. Part E will study midazolam alone and with LY3839840. The study will last up to approximately 7 weeks for parts A, C (single dose cohort), 8 weeks for parts B, D and C (multiple dose cohort), and up to 3 weeks for Part E.

ELIGIBILITY:
Inclusion Criteria:

Healthy men and women. Women may only be included if they are of nonchildbearing potential

For Part C:

• Part C of the study includes Chinese participants only. To qualify, the participants must be considered as native Chinese, defined as all the participant's biological grandparents being of Chinese origin

For Part D:

* Part D of the study includes Japanese participants only. To qualify, the participants must be first-generation Japanese, defined as the participant's biological parents, and all the participant's biological grandparents, being of exclusive Japanese descent, and being born in Japan
* Participants who are healthy as determined through medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead (electrocardiogram ECG)
* Have a body mass index (BMI) of greater than or equal to 18 to less than or equal to 35 kilograms per square meter (kg/m²). For Parts C and D: BMI greater than or equal to 18 to less than or equal to 29 kilograms per square meter (kg/m²)
* Participants who have laboratory tests within the normal reference range for the population or CRU or have results with acceptable deviations that are judged by the investigator not to be clinically significant
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Have known allergies to LY3839840, related compounds, or any components of the formulation
* Have a history or presence of multiple or severe allergies, anaphylactic reaction to prescription or nonprescription drugs, or history of significant atopy
* Have a significant history of or current rheumatologic, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (such as Cushing syndrome, hyperthyroidism, hyperaldosteronism), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational medicinal product; or of interfering with the interpretation of data
* Have had any significant infections within 3 months prior to the screening visit, or develop any of these infections before the randomization visit.
* Have received ≥1 live vaccine within 28 days of screening, or intend to during the study, or ≤28 days after the study
* Had any surgical procedure (except for minor surgery requiring local or no anesthesia and without any complications or sequelae) within 12 weeks prior to screening, or intend to during the study, or ≤28 days after the study
* Had any malignancy within the past 5 years. Exceptions: successfully treated basal cell skin carcinoma or squamous cell skin carcinoma with no evidence of recurrence or metastatic disease within the past 3 years
* Have a history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection that, in the opinion of the sponsor or investigator, poses an unacceptable risk to the participant
* Have used, or intend to use, prescription or nonprescription medication within 14 days prior to dosing (or 5 half-lives - whichever is longer)
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated in a clinical study involving an investigational product within the last 30 days of the final drug administration (or 5 half-lives - whichever is longer)
* Show evidence of active or latent TB
* Are females who are lactating or have a positive pregnancy test at screening or Day -1
* Blood donation of ≥450 mL, or participation in a clinical study that required a blood volume of ≥400 mL since the last study visit within the past 120 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more Adverse Event (s) (AEs), Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration | Baseline up to Week 8
  A summary of AEs, TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3839840 | Predose on day 1 up to 14 days post dose
  PK:Cmax of LY3839840
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3839840 | Predose on day 1 up to 14 days post dose
  PK: AUC of LY3839840
PK: AUC of Midazolam | Predose on day 1 up to 19 days post-dose
  PK: AUC of Midazolam
PK: Cmax of Midazolam | Predose on day 1 up to 19 days post-dose
  PK: Cmax of Midazolam

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - CenExel ACT, Anaheim, California
  - Fortrea Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No